CLINICAL TRIAL: NCT00006400
Title: Pediatric Hydroxyurea Phase III Clinical Trial (BABY HUG)
Brief Title: Hydroxyurea to Prevent Organ Damage in Children With Sickle Cell Anemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 89; N01HB07150 (NIH); N01HB07151 (NIH); N01HB07152 (NIH); N01HB07153 (NIH); N01HB07154 (NIH); N01HB07155 (NIH); N01HB07156 (NIH); N01HB07157 (NIH); N01HB07158 (NIH); N01HB07159 (NIH); N01HB07160 (NIH)
Record Dates: First submitted 2000-10-12; First posted 2000-10-13 (Estimated); Results first posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2011-04

CONDITIONS: Hematologic Diseases; Anemia, Sickle Cell
Keywords: Blood Diseases; Sickle Cell Anemia
MeSH Terms: conditions — Hematologic Diseases; Anemia, Sickle Cell | interventions — Hydroxyurea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hydroxyurea (Active Comparator): Participants will receive hydroxyurea.
  Interventions: Drug: Hydroxyurea
- Placebo (Placebo Comparator): Participants will receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydroxyurea — Participants will receive hydroxyurea.
  Arms: Hydroxyurea
Drug: Placebo — Participants will receive placebo.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if hydroxyurea therapy is effective in the prevention of chronic end organ damage in pediatric patients with sickle cell anemia.

DETAILED DESCRIPTION:
BACKGROUND:

In 1995, the Multicenter Study of Hydroxyurea (MSH) demonstrated that hydroxyurea is effective in decreasing the frequency of painful crises, hospitalizations for crises, acute chest syndrome, and blood transfusions by 50%. The recently completed phase II study of hydroxyurea in children (PED HUG) demonstrated that children have a response to hydroxyurea similar to that seen in adults in terms of increasing fetal hemoglobin levels and total hemoglobin, and decreasing complications associated with sickle cell anemia. In addition, this study demonstrated that the drug does not adversely affect growth and development between the ages of 5 and 15. A recently completed pilot study of hydroxyurea given to children between the ages of 6 months and 24 months demonstrated that the drug is tolerated well by small infant, and that the fetal hemoglobin switch can be forced to remain in the "on position" by hydroxyurea administration.

A Special Emphasis Panel (SEP) met on April 12, 1996 to review the results of the MSH trial and the progress to date of the PED HUG study. The SEP recommended that NHLBI undertake the BABY HUG trial.

DESIGN NARRATIVE:

BABY HUG is a randomized, double-blind, placebo-controlled study to determine if hydroxyurea can prevent the onset of chronic end organ damage in young children with sickle cell anemia. Approximately 200 children with sickle cell disease will be recruited to receive either hydroxyurea or placebo. The children will be screened at study entry for signs of abnormal brain, kidney, pulmonary, and splenic function, and developmental milestones. They will then be randomly assigned to receive either hydroxyurea or placebo and followed yearly to assess chronic end organ damage of the major organ systems. The primary endpoint will be a 50% reduction in rates of damage to the major organs with surrogate markers of organ function during follow-up in Phase II of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Majority fetal and sickle (FS or SF) hemoglobin pattern confirmed centrally by electrophoresis (screening may begin at 7 months of age)

Exclusion Criteria:

* Chronic transfusion therapy
* Cancer
* Less than 5th percentile (10th percentile for the pilot study) height, weight, or head circumference for age
* Severe developmental delay (e.g., cerebral palsy or other mental retardation, Grade III/IV intraventricular hemorrhage)
* Stroke with neurological deficit
* Surgical splenectomy
* Participating in other clinical intervention trials
* Probable or known diagnosis of Hemoglobin S-Hereditary Persistence of Fetal Hemoglobin
* Known hemoglobin S-beta plus thalassemia (hemoglobin A present)
* Any condition or chronic illness, which in the opinion of the principal investigator, makes participation unadvised or unsafe
* Inability or unwillingness to complete baseline (pre-enrollment) studies, including blood or urine specimen collection, liver-spleen scan, abdominal sonogram, neurological examination, neuropsychological testing, or transcranial Doppler ultrasound (interpretable study not required, but confirmed velocity greater than 200 cm/sec results in ineligibility)
* Previous or current treatment with hydroxyurea (HU) or another anti-sickling drug
* The following exclusion criteria are transient; patients can be re-evaluated for eligibility:

  1. Hemoglobin less than 6.0 gm/dL
  2. Reticulocyte count less than 80,000/cu mm if hemoglobin is less than 9 gm/dL
  3. Neutrophil count less than 2,000/cu mm
  4. Platelet count less than 130,000/cu mm
  5. Blood transfusion in the 2 months prior to study entry unless HbA is less than 10%
  6. ALT greater than twice the upper limit of normal
  7. Ferritin less than 10 ng/ml
  8. Serum creatinine greater than twice the upper limit of normal for age
  9. Bayley standardized mental score below 70

Ages: 9 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 193 (Actual)
Dates: Start 2000-08; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherron Jackson, MD, Principal Investigator — Medical University of South Carolina; James F. Casella, MD, Principal Investigator — Johns Hopkins University; Lori Luchtman-Jones, MD, Principal Investigator — Children's National Research Institute; Rathi V. Iyer, MD, Principal Investigator — University of Mississippi Medical Center; Scott T. Miller, MD, Principal Investigator — SUNY Health Science Center, Brooklyn; Sohail R. Rana, MD, Principal Investigator — Howard University; Zora R. Rogers, MD, Principal Investigator — University of Texas SW Medical Center; Bruce W Thompson, Ph.D., Principal Investigator — Clinical Trials and Surveys Corp; Julio Barredo, MD, Principal Investigator — University of Miami Medical Center; Winfred C. Wang, MD, Study Chair — St. Jude Children's Research Hospital; Courtney Thornburg, MD, Principal Investigator — Duke University; Thomas Howard, MD, Principal Investigator — University of Alabama at Birmingham; Lori Luck, MD, Principal Investigator — Drexel University; R. Clark Brown, MD, PhD, Principal Investigator — Emory University; Sharada Sarnaik, MD, Principal Investigator — Wayne State University
Locations (14):
- United States (14):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Howard University, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Johns Hopkins University, Baltimore, Maryland
  - Children's Hospital of Michigan/Wayne State Univ., Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - SUNY Health Science Center, Brooklyn, Brooklyn, New York
  - Duke University Medical Center, Durham, North Carolina
  - Drexel University, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - University of Texas SW Medical Center, Dallas, Texas

REFERENCES:
- [Background] Heeney MM, Whorton MR, Howard TA, Johnson CA, Ware RE. Chemical and functional analysis of hydroxyurea oral solutions. J Pediatr Hematol Oncol. 2004 Mar;26(3):179-84. doi: 10.1097/00043426-200403000-00007. PMID 15125610
- [Background] Thompson BW, Miller ST, Rogers ZR, Rees RC, Ware RE, Waclawiw MA, Iyer RV, Casella JF, Luchtman-Jones L, Rana S, Thornburg CD, Kalpatthi RV, Barredo JC, Brown RC, Sarnaik S, Howard TH, Luck L, Wang WC. The pediatric hydroxyurea phase III clinical trial (BABY HUG): challenges of study design. Pediatr Blood Cancer. 2010 Feb;54(2):250-5. doi: 10.1002/pbc.22269. PMID 19731330
- [Result] Wang WC, Ware RE, Miller ST, Iyer RV, Casella JF, Minniti CP, Rana S, Thornburg CD, Rogers ZR, Kalpatthi RV, Barredo JC, Brown RC, Sarnaik SA, Howard TH, Wynn LW, Kutlar A, Armstrong FD, Files BA, Goldsmith JC, Waclawiw MA, Huang X, Thompson BW; BABY HUG investigators. Hydroxycarbamide in very young children with sickle-cell anaemia: a multicentre, randomised, controlled trial (BABY HUG). Lancet. 2011 May 14;377(9778):1663-72. doi: 10.1016/S0140-6736(11)60355-3. PMID 21571150
- [Result] Wang WC, Pavlakis SG, Helton KJ, McKinstry RC, Casella JF, Adams RJ, Rees RC; BABY HUG Investigators. MRI abnormalities of the brain in one-year-old children with sickle cell anemia. Pediatr Blood Cancer. 2008 Nov;51(5):643-6. doi: 10.1002/pbc.21612. PMID 18478575
- [Result] Miller ST, Wang WC, Iyer R, Rana S, Lane P, Ware RE, Li D, Rees RC; BABY-HUG Investigators. Urine concentrating ability in infants with sickle cell disease: baseline data from the phase III trial of hydroxyurea (BABY HUG). Pediatr Blood Cancer. 2010 Feb;54(2):265-8. doi: 10.1002/pbc.22189. PMID 19621454
- [Result] Pavlakis SG, Rees RC, Huang X, Brown RC, Casella JF, Iyer RV, Kalpatthi R, Luden J, Miller ST, Rogers ZR, Thornburg CD, Wang WC, Adams RJ; BABY HUG Investigators. Transcranial doppler ultrasonography (TCD) in infants with sickle cell anemia: baseline data from the BABY HUG trial. Pediatr Blood Cancer. 2010 Feb;54(2):256-9. doi: 10.1002/pbc.22282. PMID 19813252
- [Result] Thornburg CD, Rogers ZR, Jeng MR, Rana SR, Iyer RV, Faughnan L, Hassen L, Marshall J, McDonald RP, Wang WC, Huang X, Rees RC; BABY HUG Investigators. Adherence to study medication and visits: data from the BABY HUG trial. Pediatr Blood Cancer. 2010 Feb;54(2):260-4. doi: 10.1002/pbc.22324. PMID 19856395
- [Result] Ware RE, Rees RC, Sarnaik SA, Iyer RV, Alvarez OA, Casella JF, Shulkin BL, Shalaby-Rana E, Strife CF, Miller JH, Lane PA, Wang WC, Miller ST; BABY HUG Investigators. Renal function in infants with sickle cell anemia: baseline data from the BABY HUG trial. J Pediatr. 2010 Jan;156(1):66-70.e1. doi: 10.1016/j.jpeds.2009.06.060. PMID 19880138
- [Result] Wynn L, Miller S, Faughnan L, Luo Z, Debenham E, Adix L, Fish B, Hustace T, Kelly T, Macdermott M, Marasciulo J, Martin B, McDuffie J, Murphy M, Rackoff B, Reed C, Seaman P, Thomas G, Wang W. Recruitment of infants with sickle cell anemia to a Phase III trial: data from the BABY HUG study. Contemp Clin Trials. 2010 Nov;31(6):558-63. doi: 10.1016/j.cct.2010.08.007. Epub 2010 Aug 24. PMID 20797449
- [Result] Rogers ZR, Wang WC, Luo Z, Iyer RV, Shalaby-Rana E, Dertinger SD, Shulkin BL, Miller JH, Files B, Lane PA, Thompson BW, Miller ST, Ware RE; BABY HUG. Biomarkers of splenic function in infants with sickle cell anemia: baseline data from the BABY HUG Trial. Blood. 2011 Mar 3;117(9):2614-7. doi: 10.1182/blood-2010-04-278747. Epub 2011 Jan 7. PMID 21217080
- [Derived] Wang WC, Oyeku SO, Luo Z, Boulet SL, Miller ST, Casella JF, Fish B, Thompson BW, Grosse SD; BABY HUG Investigators. Hydroxyurea is associated with lower costs of care of young children with sickle cell anemia. Pediatrics. 2013 Oct;132(4):677-83. doi: 10.1542/peds.2013-0333. Epub 2013 Sep 2. PMID 23999955
- [Derived] Thornburg CD, Files BA, Luo Z, Miller ST, Kalpatthi R, Iyer R, Seaman P, Lebensburger J, Alvarez O, Thompson B, Ware RE, Wang WC; BABY HUG Investigators. Impact of hydroxyurea on clinical events in the BABY HUG trial. Blood. 2012 Nov 22;120(22):4304-10; quiz 4448. doi: 10.1182/blood-2012-03-419879. Epub 2012 Aug 22. PMID 22915643
- [Derived] Alvarez O, Miller ST, Wang WC, Luo Z, McCarville MB, Schwartz GJ, Thompson B, Howard T, Iyer RV, Rana SR, Rogers ZR, Sarnaik SA, Thornburg CD, Ware RE; BABY HUG Investigators. Effect of hydroxyurea treatment on renal function parameters: results from the multi-center placebo-controlled BABY HUG clinical trial for infants with sickle cell anemia. Pediatr Blood Cancer. 2012 Oct;59(4):668-74. doi: 10.1002/pbc.24100. Epub 2012 Jan 31. PMID 22294512
- [Derived] Lebensburger JD, Miller ST, Howard TH, Casella JF, Brown RC, Lu M, Iyer RV, Sarnaik S, Rogers ZR, Wang WC; BABY HUG Investigators. Influence of severity of anemia on clinical findings in infants with sickle cell anemia: analyses from the BABY HUG study. Pediatr Blood Cancer. 2012 Oct;59(4):675-8. doi: 10.1002/pbc.24037. Epub 2011 Dec 20. PMID 22190441
- [Derived] Miller ST, Rey K, He J, Flanagan J, Fish BJ, Rogers ZR, Wang WC, Ware RE; BABY HUG Investigators. Massive accidental overdose of hydroxyurea in a young child with sickle cell anemia. Pediatr Blood Cancer. 2012 Jul 15;59(1):170-2. doi: 10.1002/pbc.23244. Epub 2011 Jul 8. PMID 21744485
- [Derived] McCarville MB, Luo Z, Huang X, Rees RC, Rogers ZR, Miller ST, Thompson B, Kalpatthi R, Wang WC; BABY HUG Investigators. Abdominal ultrasound with scintigraphic and clinical correlates in infants with sickle cell anemia: baseline data from the BABY HUG trial. AJR Am J Roentgenol. 2011 Jun;196(6):1399-404. doi: 10.2214/AJR.10.4664. PMID 21606305

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 200 patients planned; 233 patients screened; 197 patients eligible for study participation; 193 patients randomized to study treatment; 191 patients initiated study treatment
Period: Overall Study
Arm/Group | Hydroxyurea | Placebo
Started | 96 | 97
Completed | 83 | 84
Not Completed | 13 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydroxyurea | Placebo | Total
Number analyzed (Participants) | 96 | 97 | 193
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 96 | 97 | 193
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Months] | 13.57 (2.60) | 13.56 (2.74) | 13.56 (2.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 57 | 109
  Male | 44 | 40 | 84
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 94 | 87 | 181
  White | 0 | 1 | 1
  More than one race | 0 | 5 | 5
  Unknown or Not Reported | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 96 | 97 | 193

OUTCOME MEASURES:

1. Primary Outcome: Treatment Differences of the Change in Qualitative Splenic Function From Baseline
Description: Primary Endpoint: Spleen function was assessed by uptake of 99mTc sulfur colloid on liver-spleen scan before initiation of treatment (baseline) and 2 years later (exit). The results of each of the two scans were categorized as normal, functional but abnormal, or not functional by a panel of nuclear medicine specialists blinded to treatment assignment. The proportion of patients whose paired scans demonstrated a decline in splenic function was compared in the hydroxyurea versus placebo groups.
  The change in splenic function from baseline to 2 years was defined as worse if it changed from normal to decreased or absent, or decreased to absent; and not worse if it changed from decreased to decreased, normal to normal, or decreased to normal.
Time Frame: Before initiation of treatment and at 2 years
Population: Subjects who had baseline and 2 years splenic function measurements, and had baseline measurement different from absent splenic function. A total of 26 hydroxyurea and 23 placebo subjects had missing data or had absent splenic function at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxyurea | Placebo
Number analyzed (Participants) | 70 | 74
Participants
  Worse | 19 | 28
  Not worse | 51 | 46
Statistical Analysis 1: Comparison: Hydroxyurea vs Placebo; The primary analysis compared the frequency of worsening spleen function (from normal to decreased or absent, or decreased to absent) and not worsening (from decreased to decreased, normal to normal, or decreased to normal) as measured by splenic uptake on a technetium-99m (99mTc) sulfur colloid liver-spleen scan. Children with missing data or absent spleen function at baseline were excluded from the analysis (26 subjects from hydroxyurea and 23 subjects from placebo group were excluded); Test type: Superiority — The primary analysis was done using an intention-to-treat principle; p = 0.21, Fisher Exact — The spleen endpoint was to be tested at an overall alpha = 0.04. Originally there was a second primary outcome to be tested at alpha = 0.01, but this outcome was dropped

2. Secondary Outcome: Change From Baseline in the Renal Function That Was Measured by Diethylenetriaminepentaacetic Acid (DTPA) Glomerular Filtration Rate (GFR)
Description: DTPA GFR was originally a co-primary efficacy outcome for the study. Later in May 29, 2009, this measurement was discontinued because of statistical futility (an extremely small chance that the difference between treatment groups would be statistically significant for this outcome) and the small risk posed by the radiation exposure involved with performing the DTPA GFR test. Subjects who had missing data at baseline or 2 years measurement were excluded from the analysis (29 subjects from the hydroxurea, and 31 subjects from the placebo group excluded).
Time Frame: Before initiation of treatment and at 2 years
Population: Subjects who had baseline and 2 years measurements
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Hydroxyurea | Placebo
Number analyzed (Participants) | 67 | 66
mL/min/1.73m^2 | 22.56 (54.67) | 20.74 (51.07)
Statistical Analysis 1: Comparison: Hydroxyurea vs Placebo; The change from baseline to exit as measured by DTPA GFR were compared between treatment groups; Test type: Superiority; p = 0.93, ANOVA — This was originally a second primary outcome to be tested at alpha = 0.01, but was later dropped from the protocol. We analyzed the available data

3. Secondary Outcome: Change From Baseline in the Renal Function That Was Measured by Glomerular Filtration Rate (GFR) (Calculated Using Schwartz Formula)
Description: Schwartz formula used to calculate GFR is: 0.55× height (cm)/serum creatinine (mg/dL). Where height is in cm and serum creatinine is in mg/dL. Children with missing baseline or 2 years GFR were excluded from the analysis.
Time Frame: Before initiation of treatment and at 2 years
Population: All subjects who had baseline and 2 years GFR calculated using Schwartz formula (0.55× height (cm)/serum creatinine (mg/dL)).
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Hydroxyurea | Placebo
Number analyzed (Participants) | 70 | 76
mL/min/1.73m^2 | 28.65 (76.46) | 33.36 (95.85)
Statistical Analysis 1: Comparison: Hydroxyurea vs Placebo; The change from baseline to exit as measured by GFR (calculated using Shwartz formula) were compared between treatment groups; Test type: Superiority; p = 0.43, ANOVA — All secondary outcomes were tested at alpha=0.01

4. Secondary Outcome: Change From Baseline in the Renal Function That Was Measured by GFR (Calculated Using New Schwartz Formula)
Description: GFR was calculated using new Schwartz formula: 39.1× [height (cm)/serum creatinine (mg/dL)]0.516 × [1.8/cystatin C]0.294 × [30/blood urea nitrogen]0.169 × [1.099]if male × [height(m)/1.4]0.188. Children with missing baseline or 2 years GFR were excluded from the analysis.
Time Frame: Before initiation of treatment and at 2 years
Population: All subjects who had baseline and 2 years GFR calculated using the new Schwartz formula (39.1× [height (cm)/serum creatinine (mg/dL)]0.516 × [1.8/cystatin C]0.294 × [30/blood urea nitrogen]0.169 × [1.099]if male × [height(m)/1.4]0.188).
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Hydroxyurea | Placebo
Number analyzed (Participants) | 34 | 47
mL/min/1.73m^2 | 10.57 (20.78) | 14.33 (24.01)
Statistical Analysis 1: Comparison: Hydroxyurea vs Placebo; The change in GFR from baseline to exit were compared between treatment groups. GFR was calculated using new Schwartz formula; Test type: Superiority; p = 0.48, ANOVA — All secondary outcomes were to be tested at alpha = 0.01

ADVERSE EVENTS:
Time Frame: From randomization through study completion, an average of 1.93 years.
Description: The CC, NHLBI, and the DSMB continuously monitored the safety of study treatments.
  A serious adverse event(SAE) was defined as an untoward medical event that is fatal, life threatening, causes/prolongs a hospitalization, or poses a risk of permanent disability, i.e. SAE was defined as one or more of the following:
  1. Death
  2. Life-threatening events
  3. Prolonged hospitalization (greater than 7 days)
  4. Splenic sequestration crisis
  5. Stroke, TIA
  6. Acute chest syndrome
  7. ICU admissions
Groups:
- Hydroxyurea: Participants were to receive hydroxyurea.
- Placebo: Participants were to receive placebo.
Arm/Group | Hydroxyurea | Placebo
All-Cause Mortality (participants affected / at risk) | 0/96 | 0/97
Serious Adverse Events (participants affected / at risk) | 19/96 | 35/97
Other Adverse Events (participants affected / at risk) | 95/96 | 95/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxyurea (N=96) | Placebo (N=97)
Splenic Sequestration (Blood and lymphatic system disorders) | 11 (16) | 12 (17)
Acute Chest Syndrome (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 19 (28)
Acute chest syndrome (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
STROKE, WITH NEUROLOGIC DEFICIT (Nervous system disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
ACUTE OSTEOMYELITIS (Infections and infestations) | 0 (0) | 1 (1)
APLASTIC CRISIS (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
FEVER > 101.5°F(38.4°C) (General disorders) | 1 (1) | 0 (0)
SEPSIS OR MENINGITIS (Infections and infestations) | 0 (0) | 2 (2)
anemia (Hgb 6.3 - given PRBC transfusion) (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bacteremia (Infections and infestations) | 0 (0) | 1 (1)
Streptococcus pneumonieae (Infections and infestations) | 0 (0) | 1 (1)
Possible Accidental Hydroxyurea overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ABNORMAL TCD (Investigations) | 1 (1) | 3 (3)
dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
encephalopathy (indeterminate etiology) (Nervous system disorders) | 0 (0) | 1 (1)
severe obstructive sleep apnea (Nervous system disorders) | 0 (0) | 1 (1)
DVT (Vascular disorders) | 1 (1) | 0 (0)
Acute chest syndrome (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxyurea (N=96) | Placebo (N=97)
FEVER >101.5 F (38.4 C) (General disorders) | 75 (231) | 82 (272)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 83 (298) | 77 (326)
UPPER RESPIRATORY INFECTION (Respiratory, thoracic and mediastinal disorders) | 8 (12) | 14 (16)
Pain (General disorders) | 50 (131) | 62 (268)
Pain (Musculoskeletal and connective tissue disorders) | 15 (20) | 27 (49)
Pain (Gastrointestinal disorders) | 10 (13) | 15 (35)
Viral Syndrome (Infections and infestations) | 46 (69) | 46 (80)
Viral Syndrome (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (6)
Otitis Media (Infections and infestations) | 38 (80) | 48 (103)
Otitis Media (Ear and labyrinth disorders) | 11 (12) | 10 (13)
GASTROENTERITIS (Infections and infestations) | 33 (45) | 31 (47)
GASTROENTERITIS (Gastrointestinal disorders) | 7 (10) | 3 (3)
SPLENOMEGALY (Blood and lymphatic system disorders) | 32 (105) | 35 (84)
CONSTIPATION (Gastrointestinal disorders) | 16 (23) | 33 (65)
SKIN INFECTION, FUNGAL (Infections and infestations) | 15 (21) | 13 (14)
SKIN INFECTION, FUNGAL (Skin and subcutaneous tissue disorders) | 1 (1) | 6 (7)
DACTYLITIS (Musculoskeletal and connective tissue disorders) | 14 (23) | 43 (123)
SKIN INFECTION, BACTERIAL (Infections and infestations) | 5 (5) | 9 (14)
Pneumonia (Infections and infestations) | 11 (14) | 21 (28)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 11 (12)
Eczema (Skin and subcutaneous tissue disorders) | 11 (15) | 12 (18)
Rash (Skin and subcutaneous tissue disorders) | 21 (25) | 29 (43)
Diarrhea (Gastrointestinal disorders) | 12 (15) | 14 (14)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 15 (21)
CONJUNCTIVITIS (Infections and infestations) | 16 (18) | 13 (16)
Emesis (Gastrointestinal disorders) | 7 (9) | 9 (11)
URI (Infections and infestations) | 2 (3) | 6 (9)
Insect Bites (Injury, poisoning and procedural complications) | 12 (15) | 15 (22)
Vomiting (Gastrointestinal disorders) | 11 (13) | 14 (15)
Bronchitis (Infections and infestations) | 4 (7) | 6 (7)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 8 (11) | 3 (4)
Urinary Tract Infection (Infections and infestations) | 5 (7) | 11 (13)
Low Grade Fever (<101.5) (General disorders) | 9 (12) | 14 (18)
Reactive Airway Disease (Respiratory, thoracic and mediastinal disorders) | 5 (9) | 9 (13)
RHINORRHEA (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 11 (15)
PHARYNGITIS (Infections and infestations) | 7 (7) | 5 (6)
SINUSITIS (Infections and infestations) | 3 (3) | 6 (6)
Asthma (Respiratory, thoracic and mediastinal disorders) | 8 (13) | 6 (9)
Diaper DERMATITIS (Skin and subcutaneous tissue disorders) | 7 (7) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2009-08-09): https://cdn.clinicaltrials.gov/large-docs/00/NCT00006400/Prot_SAP_000.pdf
  • Informed Consent Form (2006-10-16): https://cdn.clinicaltrials.gov/large-docs/00/NCT00006400/ICF_001.pdf